CLINICAL TRIAL: NCT07230561
Title: The Efficacy of Structured Early Mobilization Training in Patients After Coronary Artery Bypass Surgery: A Randomized Controlled Trial
Brief Title: Early Mobilization After CABG Surgery
Acronym: EMAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ta-Chung Chao (Other)
Collaborators: Far Eastern Memorial Hospital (Other); Tri-Service General Hospital (Other)
Responsible Party: Sponsor-Investigator, Ta-Chung Chao, Principal Investigator, National Defense Medical Center, Taiwan
Organization: National Defense Medical Center, Taiwan (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 113105-F; FEMH-2024-C-094 (Other Grant/Funding Number: Far Eastern Medical Foundation Far Eastern Memorial Hospital)
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease; Coronary Artery Bypass
Keywords: Cardiorespiratory Fitness; Coronary Artery Bypass; Early Mobilization; Postoperative Care; Quality of Life; Randomized Controlled Trial; Sarcopenia
MeSH Terms: conditions — Coronary Artery Disease; Sarcopenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Participants received standard hospital nursing care PLUS supervised, structured early mobilization training. The protocol was developed by integrating Phase 1 cardiac rehabilitation guidelines with an expert consensus approach from a multidisciplinary team. The intervention began within 24 hours postoperatively, was conducted for 5 days, twice daily, 30 min/session. Sessions included a 5-min warm-up (active/passive ROM), a 20-min main training (FITT principle: Intensity at resting heart rate + 20 bpm, max 120 bpm; Type: inspiratory muscle training, ROM, stationary cycling or bedside ambulation, resistance training), and a 5-min cool-down.
  Interventions: Behavioral: Structured Early Mobilization Training; Other: Standard Hospital Nursing Care
- Comparison Group (Active Comparator): Participants received standard hospital nursing care only. This included physiological monitoring, medication counseling, psychological support, disease-specific health education, instruction on the use of an incentive spirometer, and education on the importance and methods of rehabilitation.
  Interventions: Other: Standard Hospital Nursing Care

INTERVENTIONS:
Behavioral: Structured Early Mobilization Training — The training protocol was developed by integrating Phase 1 cardiac rehabilitation guidelines with an expert consensus approach from a multidisciplinary team. The intervention began within 24 hours postoperatively, was conducted for 5 days, twice daily, 30 min/session. Sessions included a 5-min warm-up (active/passive ROM), a 20-min main training (FITT principle: Intensity at resting heart rate + 20 bpm, max 120 bpm; Type: inspiratory muscle training, ROM, stationary cycling or bedside ambulation, resistance training), and a 5-min cool-down.
  Arms: Exercise Group
Other: Standard Hospital Nursing Care — The standard hospital nursing care included physiological monitoring, medication counseling, psychological support, disease-specific health education, instruction on the use of an incentive spirometer, and education on the importance and methods of rehabilitation.

SUMMARY:
The goal of this clinical trial is to learn if a structured early exercise program can help patients recover better in people who have just had coronary artery bypass surgery. The main questions it aims to answer are:

* Does this early exercise improve fitness and walking ability?
* Does it reduce the risk of muscle weakness (sarcopenia) after surgery?
* Does it improve patients' quality of life?
* Does it reduce feelings of anxiety and depression? Researchers will compare the group receiving the structured early exercise program (plus standard hospital care) to the group receiving standard hospital care only to see if the early exercise program leads to better and faster recovery.

Participants in the exercise group will:

* Start supervised exercise sessions within 24 hours after their surgery.
* Perform these sessions twice a day for 30 minutes each, for 5 days.
* The exercises include warm-ups, breathing exercises, walking or stationary cycling, and light resistance training.

ELIGIBILITY:
Inclusion Criteria:

* age between 40 and 85 years;
* undergoing first-time CABG surgery;
* no diagnosed psychiatric disorders or musculoskeletal diseases and did not require any assistive mobility devices;
* ability to communicate in Mandarin or Taiwanese;
* agreed to participate and provided written informed consent after receiving a comprehensive explanation of this trial.

Exclusion Criteria:

* preoperative use of continuous 24-hour nitroglycerin infusion or inotropic agents;
* undergoing emergency cardiac surgery or requiring admission to the intensive care unit preoperatively;
* occurrence of major intraoperative complications (e.g., major hemorrhage, stroke, requirement for resuscitation, or severe delirium).

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Cardiorespiratory Fitness | Baseline (preoperative at admission), Postoperative Day 6, Postoperative Day 14
  Assessed by the 6-minute walk test (6MWT). Total distance (in meters) walked along a 30-meter flat corridor in six minutes.
Change in Sarcopenia Risk Classification | Baseline (preoperative at admission), Postoperative Day 6, Postoperative Day 14
  Assessed using the Strength, Assistance with walking, Rising from a chair, Climbing stairs, and Falls (SARC-F) questionnaire. The total score ranges from 0 to 10. Higher scores indicate a greater risk of sarcopenia (worse outcome). Classified as "at risk" (SARC-F total score more than or equal to 4 points) or "not at risk".
Change in Strength, Assistance with walking, Rising from a chair, Climbing stairs, and Falls (SARC-F) Total Score | Baseline (preoperative at admission), Postoperative Day 6, Postoperative Day 14
  Assessed using the Strength, Assistance with walking, Rising from a chair, Climbing stairs, and Falls (SARC-F) questionnaire. The total score ranges from 0 to 10. Higher scores indicate a greater risk of sarcopenia (worse outcome).
Change in Muscle Strength (Left Handgrip) | Baseline (preoperative at admission), Postoperative Day 6, Postoperative Day 14
  Assessed by maximal handgrip strength (in kg) using a hydraulic dynamometer.
Change in Muscle Strength (Right Handgrip) | Baseline (preoperative at admission), Postoperative Day 6, Postoperative Day 14
  Assessed by maximal handgrip strength (in kg) using a hydraulic dynamometer.
Change in Physical Performance (5-Times Sit-to-Stand Test) | Baseline (preoperative at admission), Postoperative Day 6, Postoperative Day 14
  Time (in seconds) taken to stand and sit five times from a chair with arms crossed.
Change in Muscle Mass Proxy (Left Calf Circumference) | Baseline (preoperative at admission), Postoperative Day 6, Postoperative Day 14
  Maximum circumference (in cm) at the widest part of the calf while seated.
Change in Muscle Mass Proxy (Right Calf Circumference) | Baseline (preoperative at admission), Postoperative Day 6, Postoperative Day 14
  Maximum circumference (in cm) at the widest part of the calf while seated.
Change in Quality of Life | Baseline (preoperative at admission), Postoperative Day 6, Postoperative Day 14
  Assessed using the EuroQol 5-Dimension 3-Level (EQ-5D-3L) questionnaire. The index score typically ranges from 0 to 1.00. Higher scores indicate a better quality of life (better outcome), with 1.00 representing perfect health and 0 representing death.
Change in Self-Rated Health | Baseline (preoperative at admission), Postoperative Day 6, Postoperative Day 14
  Assessed using the EuroQol visual analogue scale (EQ-VAS). Scale 0 (worst imaginable) to 100 (best imaginable).
Change in Mood (Anxiety) | Baseline (preoperative at admission), Postoperative Day 6, Postoperative Day 14
  Assessed using the Hospital Anxiety and Depression Scale (HADS) Anxiety subscale. Score ranges from 0 to 21. Higher scores indicate higher levels of anxiety (worse outcome).
Change in Mood (Depression) | Baseline (preoperative at admission), Postoperative Day 6, Postoperative Day 14
  Assessed using the Hospital Anxiety and Depression Scale (HADS) Depression subscale. Score ranges from 0 to 21. Higher scores indicate higher levels of depression (worse outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Medical Foundation Far Eastern Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in the final publication will be made available. The study protocol will also be available.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available beginning 6 months after the publication of the primary manuscript and will remain available for 5 years.
Access Criteria: Data access will be granted to qualified academic researchers for legitimate research purposes, such as re-analysis or meta-analysis. Researchers must submit a methodologically sound proposal to the corresponding author. Upon approval by the principal investigators and the Institutional Review Board, and contingent upon the terms of the original informed consent, de-identified Individual Participant Data that underlie the results reported in the final publication (including main dataset and analytic code) will be shared. A signed data-use agreement will be required prior to data release to ensure participant confidentiality.